CLINICAL TRIAL: NCT02592538
Title: Endobiliary Radiofrequency Ablation With S-1 in Patients With Unresectable Cholangiocarcinoma: A Prospective Randomized Trial With Open Label Control
Brief Title: Endobiliary Radiofrequency Ablation With S-1 for Unresectable Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Deputy irector, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-001-003
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Cholangiocarcinoma
Keywords: Biliary duct carcinoma;; radiofrequency ablation; S-1
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiofrequency Ablation; S 1 (combination); Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA+stent+S-1 (Experimental): Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the biliary malignancy. Patients will receive endobiliary radiofrequency ablation ( RFA) followed by plastic stent(s) placement, and be treated with S-1 began within 1 month after RFA.
  Interventions: Device: radiofrequency ablation; Drug: S-1; Device: Stent
- RFA+stent (Placebo Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the biliary malignancy. Patients will only receive endobiliary radiofrequency ablation ( RFA) followed by plastic stent(s) placement
  Interventions: Device: radiofrequency ablation; Device: Stent

INTERVENTIONS:
Device: radiofrequency ablation — All patients underwent biliary sphincterotomy. Cholangiogram was performed to confirm stricture location, length and diameter. The Habib Endo HPB (Hepatobiliary) probe (EMcision, HitchinHerts, UK) was then advanced over a wire at the level of the biliary stricture and ablation using ERBE generator set at 7-10 watts for a time period of 90-120 s was conducted. A 1- to 2-min resting period after energy delivery was allowed before moving the catheter along the length of the stricture to ablate the rest of the stricture.
Drug: S-1 — In the RFA plus S-1 group, treatment with S-1 began within 1 month after RFA. Based on the patient's body surface area, S-1 was administered as follows: when the level of total bilirubin was less than 2 mg/dl. Based on the body surface area, S-1 was administered if <1.25 m2, 80 mg/day; if 1.25-1.5 m2, 100 mg/day; if≥1.5 m2, 120 mg/day. S-1 was administered orally twice daily for 14 days, followed by 7 days without treatment.
  Other Names: oral fluoropyrimidine
  Arms: RFA+stent+S-1
Device: Stent — Plastic stent(s) were placed after RFA depending on the location of the malignant obstruction

SUMMARY:
Endobiliary radiofrequency ablation (RFA) with biliary stent has been reported to be a beneficial treatment option for palliation of malignant biliary strictures. RFA uses a high-frequency alternating current to generate heat and achieve coagulative necrosis when in contact with tissue. Within the bile duct, RFA appears to be safe and may result in decreased tumor ingrowth. However, most of therapeutic effects were expected to delay bile duct obstruction rather than to decrease the tumor. Recently orally available chemotherapeutic agent, S-1, an oral fluoropyrimidine, was reported as effective in patients with bile duct adenocarcinoma. To date, little is known about the role of the addition of systemic chemotherapy to RFA for cholangiocarcinoma. The aim of this study is to evaluate the combined effect of RFA and S-1 in patients with unresectable cholangiocarcinoma.

DETAILED DESCRIPTION:
Over 60 % of common bile duct (CBD) obstructions are due to malignancy, and the majority of neoplasms are unresectable at the time of diagnosis. Biliary drainage with placement of metal or plastic stents for palliation is the therapy of choice in this set of patients.

Radiofrequency ablation (RFA) is well established method for treatment of some solid tumors, like liver cancer, lung cancer, etc. Recently, an endoscopically applicable radiofrequency probe, HabibTM EndoHBP catheter, was approved for clinical use. RFA uses a high-frequency alternating current to generate heat and achieve coagulative necrosis when in contact with tissue. Many studies showed RFA with biliary stent was a beneficial treatment option for palliation of malignant biliary strictures. However, most of therapeutic effects were expected to delay bile duct obstruction rather than to decrease the tumor. Recently orally available chemotherapeutic agent, S-1, an oral fluoropyrimidine, was reported as effective in patients with bile duct adenocarcinoma. To date, little is known about the role of the addition of systemic chemotherapy to RFA for cholangiocarcinoma.

The aim of this study is to conduct a randomised, controlled, clinical trial to compare the effect of S-1 plus RFA with stent with RFA with stent in patients with unresectable cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Obtention of a written informed consent.
* Patient over 18.
* Patient with histologically proved cholangiocarcinoma ; histologic diagnosis must be proved by biliary brushing, bile cytology, endobiliary biopsy under Spyglass, or by EUS-FNA.
* Patient with Karnofsky score ≥ 50 %
* Patient capable of fill in the quality of life questionnaire.

Exclusion Criteria:

* No written informed consent.
* Patients under or already treated by radiotherapy or chemotherapy treatment for cholangiocarcinoma.
* Patients with porphyria or hypersensibility to porphyrins.
* Pregnant, parturient or breastfeeding women.
* Patient under 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
survival time | two years
  Compare overall survival time in patients with unresectable cholangiocarcinoma treated with RFA combined with or without S-1

SECONDARY OUTCOMES:
adverse events | two years
  Number of participants with adverse events; type, frequency and intensity of adverse events
frequency of repeat RFA | two years
the frequency of cholangitis | two years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laquiere A, Boustiere C, Leblanc S, Penaranda G, Desilets E, Prat F. Safety and feasibility of endoscopic biliary radiofrequency ablation treatment of extrahepatic cholangiocarcinoma. Surg Endosc. 2016 Mar;30(3):1242-8. doi: 10.1007/s00464-015-4322-7. Epub 2015 Jul 11. PMID 26162420
- [Background] Butros SR, Shenoy-Bhangle A, Mueller PR, Arellano RS. Radiofrequency ablation of intrahepatic cholangiocarcinoma: feasability, local tumor control, and long-term outcome. Clin Imaging. 2014 Jul-Aug;38(4):490-494. doi: 10.1016/j.clinimag.2014.01.013. Epub 2014 Feb 7. PMID 24637151
- [Background] Strand DS, Cosgrove ND, Patrie JT, Cox DG, Bauer TW, Adams RB, Mann JA, Sauer BG, Shami VM, Wang AY. ERCP-directed radiofrequency ablation and photodynamic therapy are associated with comparable survival in the treatment of unresectable cholangiocarcinoma. Gastrointest Endosc. 2014 Nov;80(5):794-804. doi: 10.1016/j.gie.2014.02.1030. Epub 2014 May 15. PMID 24836747
- [Derived] Yang J, Wang J, Zhou H, Wang Y, Huang H, Jin H, Lou Q, Shah RJ, Zhang X. Endoscopic radiofrequency ablation plus a novel oral 5-fluorouracil compound versus radiofrequency ablation alone for unresectable extrahepatic cholangiocarcinoma. Gastrointest Endosc. 2020 Dec;92(6):1204-1212.e1. doi: 10.1016/j.gie.2020.04.075. Epub 2020 May 11. PMID 32437711
- [Derived] Yang J, Wang J, Zhou H, Zhou Y, Wang Y, Jin H, Lou Q, Zhang X. Efficacy and safety of endoscopic radiofrequency ablation for unresectable extrahepatic cholangiocarcinoma: a randomized trial. Endoscopy. 2018 Aug;50(8):751-760. doi: 10.1055/s-0043-124870. Epub 2018 Jan 17. PMID 29342492